CLINICAL TRIAL: NCT02180048
Title: "The Effects of Caffeine on Overactive Bladder Symptoms and Mental Health in Postmenopausal Women"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5130411
Record Dates: First submitted 2014-06-27; First posted 2014-07-02 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Overactive Bladder; Caffeine; Menopause
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 400 mg of caffeine/day (Two 200mg pills/day) (Active Comparator): One phase of treatment will have participants consume two 200 mg-caffeine pills day (total of 400 mg of caffeine/ d) for 7 days.
  Interventions: Dietary Supplement: 400 mg of caffeine/day (Two 200mg pills/day)
- 200 mg of caffeine/day (One 200mg pill and one placebo pill) (Active Comparator): This arm will receive one 200 mg caffeine pill and one sugar pill (placebo pill)
  Interventions: Dietary Supplement: 200 mg of caffeine/day (One 200mg pill and one placebo pill)
- Two placebo pills/day (Placebo Comparator): This arm will have participants consume two placebo pills each day.
  Interventions: Dietary Supplement: Two placebo pills/day

INTERVENTIONS:
Dietary Supplement: 400 mg of caffeine/day (Two 200mg pills/day) — One phase of treatment will have participants consume two 200 mg-caffeine pills day (total of 400 mg of caffeine/ d) for 7 days.
  Arms: 400 mg of caffeine/day (Two 200mg pills/day)
Dietary Supplement: 200 mg of caffeine/day (One 200mg pill and one placebo pill) — This arm will receive one 200 mg caffeine pill and one sugar pill (placebo pill)
  Arms: 200 mg of caffeine/day (One 200mg pill and one placebo pill)
Dietary Supplement: Two placebo pills/day — This arm will have participants consume two placebo pills each day.
  Arms: Two placebo pills/day

SUMMARY:
The purpose of this study is to observe effects of caffeine on overactive bladder symptoms and wellbeing. This study looks at whether caffeine has bad effects on urinary symptoms or if lower doses of caffeine decrease the effects.

The study will propose the following hypothesis:

1. The voiding and mental health symptoms will be greatest in the high dose treatment and lowest in the placebo treatment.
2. The low dose treatment will produce more voiding and mental health symptoms than the placebo treatment.
3. Voiding and mental health symptoms will be mediated by hydration status of the patient which will be assessed using a Tanita Scale.

DETAILED DESCRIPTION:
Subjects will be exposed to 200 mg and 400 mg caffeine pills and placebo pills (free of caffeine). During each treatment period, participants will be required to avoid caffeine (except for the caffeine within the given treatment). The study is staged into 3 phases, which will last for 7 days each. After enrollment, participants will be asked to refrain from consuming any substances containing caffeine during the 21 days of treatment. Instead of coffee or other caffeine items, they will be exposed to caffeine in pill form. Participants will complete each treatment in a random, cross over blinded fashion. One phase of treatment will have participants consume two 200 mg-caffeine pills a day (total of 400 mg of caffeine/day), a second treatment will have participants consume one 200 mg-caffeine pill and one placebo pill a day. And the final treatment will have participants consume two placebo pills each day. Treatment phases will be assigned randomly to each participant. The participant will not know which phase they are receiving.

Prior to the treatment, the participant will be asked to fill out a detailed diet log of her eating and drinking habits. Participants will also be asked a series of questions on a survey related to bladder symptoms and mental health periodically throughout the study. It will take about 30 minutes of their time to answer the questionnaires at individual time points.

During the 21 days of the study period participants will be asked to self-monitor fluid intake and note any major changes of fluid intake compared to the initial intake log. They will be asked to conduct a 24-hour voiding and defecation log at two different time points within each treatment phase as well as prior to the study. 24-hour urine will be collected during each treatment phase at two different time points as well as prior to the study. Participants weight and lean body mass will be assessed in clinic using a Tanita scale at two times within each treatment phase and one time prior to the study

ELIGIBILITY:
Inclusion Criteria:

* Low to moderate coffee drinkers (between 1-3 cups/day, or 50-450mg caffeine/d)
* Able to communicate and read in English
* 58 years of age or older
* Post-menopausal

Exclusion Criteria:

* Excessive coffee drinkers (>450 mg/d)
* Individual who do not regularly consume caffeine
* Uncontrolled hypertension
* Vaginal pain
* Chronic pelvic pain/ Interstitial cystitis
* Pre- or perimenopausal

Min Age: 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-07; Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Change in voiding symptoms | Voiding symptoms surveys will be completed 6 times throughout the 21-day trial, in addition to a baseline measurement pre-trial.
  Voiding symptoms will be measured through a composite of self-reported surveys. These surveys are the King's Health Questionnaire, Urinary Distress Inventory, Overactive Bladder Symptom Score, Overactive Bladder Questionnaire.
Change in mental health | Mental health symptoms will be measured 6 times throughout the 21-day trial, as well as a baseline measure one time pre-trial.
  Mental health symptoms will be measured through a composite of self-reported surveys. These surveys are the Insomnia Severity Index, Stress Quiz, Beck Anxiety Index, Beck Depression Inventory, The Positive and Negative Affect Scales, Rosenberg Self-Esteem Scale, and the International Physical Activity Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Staack, MD, Principal Investigator — Loma Linda University, Urology Medical Group, Inc.
Locations (1):
- Department of Urology, Loma Linda University, Loma Linda, California, United States

REFERENCES:
- [Derived] Staack A, Distelberg B, Moldovan C, Belay RE, Sabate J. The Impact of Caffeine Intake on Mental Health Symptoms in Postmenopausal Females with Overactive Bladder Symptoms: A Randomized, Double-Blind, Placebo-Controlled Trial. J Womens Health (Larchmt). 2022 Jun;31(6):819-825. doi: 10.1089/jwh.2021.0467. Epub 2022 Apr 1. PMID 35363563